CLINICAL TRIAL: NCT02462681
Title: Ketamine as Adjunctive Analgesic With Bupivacaine in Paravertebral Analgesia for Breast Cancer Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, lecturer of anesthesia,ICU and pain relief, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 211
Record Dates: First submitted 2015-05-30; First posted 2015-06-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Acute Pain; Chronic Pain
Keywords: ketamine; adjuvant; paravertebral block
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- bupivacaine group in paravertebral block (Active Comparator): patients will be received 20 ml of bupivacaine 0.25% paravertebrally, divided into 3-4 ml in each level
  Interventions: Drug: paravertebral block
- bupivacaine + 0.5 mg/kg ketamine group in paravertebral block (Active Comparator): patients will be received 20 ml of bupivacaine 0.25% + 0.5 mg/kg ketamine paravertebrally divide into 3-4 ml in each level
  Interventions: Drug: paravertebral block
- bupivacaine + 1 mg/kg ketamine group in paravertebral block (Active Comparator): patients will be received 20 ml of bupivacaine 0.25% + 1mg/kg ketamine paravertebrally divide into 3-4 ml in each level
  Interventions: Drug: paravertebral block

INTERVENTIONS:
Drug: paravertebral block — Thoracic paravertebral blocks will be performed as described by Moore and Katz. Intradermal lidocaine will be used at the site of the needle insertion. The superior aspect of the spinous processes of T1- T6 will be marked. The skin entry points will 3 cm laterals to the marks. A 22- gauge quincke spinal needle attach to extension tubing to a syringe containing study drugs will be used. The needle will be inserted perpendicular to the skin for a distance of 2 to 4 cm until the transverse process will contact. The needle will be withdrawn and walk cephalad off the transverse process and advance for a further 1.5 to 2 cm.
  Other Names: ketamine hydrochloride

SUMMARY:
This study aims to investigate the safety and the analgesic efficacy of adding Ketamine to bupivacaine 0.25% in thoracic PVB in patients undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
Breast cancer is perhaps the most common cancer in women that requires frequent surgical intervention. Nearly 40% of post-operative breast surgery patients experience significant acute post-operative pain, with a pain score above five reflecting inadequacy of conventional pain management. Most of the responses of the human body to post-surgical pain have been proven to be detrimental to the patient's homeostasis and recovery. Moreover, the incidence of chronic postoperative pain in breast surgery patients is as high as 50% and inadequate analgesia is considered as an independent risk factor. Hence, a number of therapeutic measures have been accepted as a part of the "multi-modal" approach to post-operative pain control. Thoracic Paravertebral Block (PVB) is used for pain relief after thoracotomy , and mastectomy. PVB can provide profound, long lasting sensory differentiation. The resulting greater attenuation of surgical stress response may translate into reduced inotropic stimulation of the heart. Additionally, unlike general anesthesia, PVB can provide superior postoperative analgesia, less nausea and vomiting, shorter recovery time; require fewer analgesic, earlier mobilization, and earlier home readiness for discharge. The use of PVB in patients undergoing ambulatory breast surgery has cost-saving potential. There is little systematic research on the efficacy and tolerability of the addition of adjunctive analgesic agent in paravertebral analgesia. The addition of adjunctive analgesics, such as fentanyl and clonidine to local anesthetics has been shown to enhance the quality and duration of sensory neural blockade, and decrease the dose of local anesthetic and supplemental analgesia .

Ketamine is an anaesthetic agent with potent analgesic properties. Its mode of action includes noncompetitive antagonism at N-methyl d-aspartate (NMDA) receptors and a local anaesthetic effect. ketamine has been extensively used through epidural and caudal routes with variable results.It possesses some definite advantages over the conventional local anaesthetic agents as it stimulates cardiovascular system and respiratory system.The advantages of ketamine include a good analgesic effect, cardio vascular stability in a hypotensive state, bronchodilatation in asthmatics, and the absence of awareness. Disadvantages include increased heart rate and blood pressure, emergence phenomenon, laryngospasm and apnea, increases in intracranial and intraocular pressure, and the lack of visceral anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for elective modified radical mastectomy with axillary dissection will be enrolled in the study

Exclusion Criteria:

* patients with a known allergy to the study drugs
* patients with bleeding diathesis
* patients with infection at the site of injection
* patients with central neuropathy
* patients with liver impairment
* patients with renal impairment
* drugs or alcohol abusers
* patients with psychiatric illnesses

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
changes in pain intensity score from baseline | at 2,4,6,12,24,36and 48 hour postoperatively
  Visual analogue scale (VAS) Scored from 0-10 (where 0= no pain and 10= the worst pain imaginable) as it measured as VAS at rest (VAS.R) and during movement or ipsilateral arm abduction (VAS.M)

SECONDARY OUTCOMES:
side effect | 2,4,6,12,24,36and 48 hour postoperatively.
  nausea, vomiting, hypotension, bradycardia, sedation, dizziness and nystagmus will recorded and treated also postoperative complications of the block such as accidental pneumothorax and vascular puncture will be recorded and treated
chronic neuropathic pain | 1st,2nd and 3rd postoperative months
  (Douleur Neuropathique 4 questions) (DN4) questionnaire will be used for assessment of development of neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: Sahar A. Mohamed, MD, Principal Investigator — Lecturer of anesthesia, ICU and pain management- South Egypt Cancer Institute- Assuit University
Locations (1):
- Assiut University, Asyut, Egypt